CLINICAL TRIAL: NCT07135011
Title: Adaptive Study to Assess the Initial Safety and Functioning of the Minimally Invasive Gluteal Augmentation Procedure and Its Devices in Participants Undergoing Primary Gluteal Enhancement
Brief Title: Adaptive Study to Assess the Safety and Functioning of Motiva Devices on Minimally Invasive Gluteal Augmentation
Acronym: GEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Establishment Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLINP-01017
Record Dates: First submitted 2024-12-02; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Device Safety
Keywords: Equipment safety; Buttock augmentation

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, adaptive, interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safety and performance of medical devices (Experimental): 120 participants will undergo primary gluteal enhancement procedures utilizing the Ergonomix2® Diamond®, Motiva Injector®, Motiva® Inflatable Balloon, Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator devices.
  Interventions: Device: Primary gluteal enhancement

INTERVENTIONS:
Device: Primary gluteal enhancement — 120 participants will undergo primary buttock enhancement procedures utilizing the Ergonomix2® Diamond®, Motiva Injector®, Motiva® Inflatable Balloon, Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator devices.

SUMMARY:
The objective of this clinical trial is to assess the initial performance and safety of Motiva® Ergonomix2® Diamond®, Motiva Injector®, Motiva® Inflatable Balloon, Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator utilized in a minimally invasive gluteal augmentation procedure, involving 120 healthy female participants.

The main questions it aims to answer are:

* Are the main side effects and complications experienced by participants who underwent a minimally invasive buttock enhancement procedure with Motiva Ergonomix2® Diamond®, the Motiva Injector®, the Motiva® Inflatable Balloon, the Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator adequately characterized?
* Can the Motiva Injector®, Motiva® Inflatable Balloon, the Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator be successfully utilized, and are any failures in the process detected?
* Does the Motiva® GEM Channel Separator effectively perform tissue dissection procedures without experiencing operational dysfunctions?
* Are both the surgeon and the participant satisfied with the procedure outcomes?
* Is the proper functioning of the Zen microtransponder verified? Participants will undergo a minimally invasive buttock enhancement procedure using the Ergonomix2® Diamond®, the Motiva Injector®, the Motiva® Inflatable Balloon, the Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator, and have a follow-up of 24 months to see the results.

DETAILED DESCRIPTION:
This is a prospective, open-label, interventional study lasting 24 months, aimed at evaluating the safety and performance of Motiva® Ergonomix2® Diamond®, Motiva Injector®, Motiva® Inflatable Balloon, Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator utilized in a minimally invasive gluteal augmentation procedure.

The devices included in this study are indicated for use in the chest area. According to an ongoing study, their safety and performance have been demonstrated. It is not expected that the off-label use of Ergonomix2® Diamond®, Motiva Injector®, Motiva® Inflatable Balloon, Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator in the gluteal area will increase any risks or potential harm to the participants. On the contrary, the minimally invasive procedure is expected to provide more positive and safer outcomes.

This study has been designed as an adaptive study since the devices to be used are not indicated for use in the gluteal area. This allows for careful evaluation of real-time clinical data to make decisions regarding clinical development. This study will consist of two stages: the feasibility stage and the pivotal stage.

It involves the decision to progress participant recruitment from the feasibility phase to the pivotal phase, as long as there are no unknown complications, serious incidents, or incidents not previously described in available literature. A pre-planned interim analysis will be conducted every 6 months. It will analyze enrolled participants, their complications, and satisfaction. The collected data will be considered to decide transition stages.

The scope of the adaptive design is to combine these two stages of clinical development to:

* Maximize trial information
* Shorten development timelines
* Reduce risk for study participants and the sponsor
* Regulatory advantages

For this study, 120 women will be recruited according to the study's requirements from different countries in Latin America to undergo a minimally invasive gluteal enhancement procedure using Ergonomix2® Diamond®, Motiva Injector®, Motiva® Inflatable Balloon, Motiva® Reusable Channel Dissector, and Motiva® GEM Channel Separator. The study period will last up to 24 months, and recruitment is expected to last up to six months.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women, aged 18 years or older.
* Participants without prior buttock augmentation or biopolymer injections in the buttocks.
* Participants classified as ASA class I and II according to the American Society of Anesthesiologists (ASA) classification system for estimating risk.
* Participants seeking buttock enhancement, aiming to simply restore the aesthetic curvature of the back.
* Body mass index between 18.5 and 28.
* Adequate tissue available to cover the implant(s).
* Willingness to comply with all study requirements and agree to attend all required follow-up visits.
* Agreement to return the device to the sponsor in case of explantation.

Exclusion Criteria:

* Women with massive weight loss.
* Buttock ptosis or poor skin quality.
* Inadequate tissue (e.g., due to radiation damage, ulceration, compromised vascularization, history of compromised healing).
* Current pregnancy.
* History of abscesses or infections in the buttock area.
* History of sensitivity to silicone.
* Any medical condition such as underweight or obesity according to inclusion criteria, diabetes, autoimmune disease, or severe chronic pulmonary or cardiovascular disease resulting in excessively high surgical risk and significant postoperative complications.
* History of psychological characteristics that are unrealistic or unreasonable given the risks associated with the surgical procedure.
* Use of any medication that, according to the investigator's experience, may pose a higher risk of complications or interfere with wound healing capacity, such as corticosteroid treatment or blood-thinning medications (e.g., concomitant treatment with warfarin).
* Participants who do not reside in the Great Metropolitan Area of Costa Rica, which makes it difficult for them to attend follow-up visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Safety e:valuation | 24 months
  Safety will be assessed through the cumulative incidence (number of cases) of adverse events during surgery and the follow-up period. The severity and duration of all complications (rate of procedure-related adverse events/device-related adverse events) will be included. Safety will be evaluated through a survival analysis.
Primary Performance Evaluation | 24 months
  The performance of the devices will be evaluated as successful in all cases of buttock enhancement where there is no device malfunction. All assessment criteria must be analyzed per participant and per buttock. A 90% confidence interval will be obtained for each parameter when applied.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Ortiz Barboza, MD, Principal Investigator — Principal Investigator
Locations (1):
- Establishment Labs, Alajuela, Provincia de San José, Costa Rica